CLINICAL TRIAL: NCT05384002
Title: An AI Platform Integrating Imaging Data and Models, Supporting Precision Care Through Prostate Cancer's Continuum
Status: Completed | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Collaborators: Fundacao Champalimaud (Other); Stichting Katholieke Universiteit (Other); Fundacion Para La Investigacion Hospital La Fe (Other); University of Pisa (Other); Institut Paoli-Calmettes (Other); Hacettepe University (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); JCC DIAGNOSTIC IMAGING (Unknown); National Cancer Institute (NCI) (NIH); Agios Savas (Unknown); Royal Marsden NHS Foundation Trust (Other); QS INSTITUTO DE INVESTIGACION E INNOVACION SL (Unknown); IDRYMA TECHNOLOGIAS KAI EREVNAS (Unknown); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); THE GENERAL HOSPITAL CORPORATION (Unknown); BIOTRONICS 3D LIMITED (Unknown); Advantis Medical Imaging (Unknown); QUIBIM SOCIEDAD LIMITADA (Unknown); University of Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: ProCAncer-I; NCT05380518 (obsolete NCT alias)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic; Prostate Cancer Recurrent; Prostate Cancer Aggressiveness
Keywords: prostate cancer; repository; open image space; annotated and under donorship images; quality of image providers; cloud infrastructure; tools to build AI applications; advanced AI techniques
MeSH Terms: conditions — Prostatic Neoplasms; Prostate Cancer, Hereditary, 7 | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective (training model)
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Prospective (validation model)
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Patients who underwent MRI with confirmed pathology data (either biopsy or prostatectomy)

SUMMARY:
In Europe, prostate cancer (PCa) is the second most frequent type of cancer in men and the third most lethal. Current clinical practices, often leading to overdiagnosis and overtreatment of indolent tumors, suffer from lack of precision calling for advanced AI models to go beyond SoA by deciphering non-intuitive, high-level medical image patterns and increase performance in discriminating indolent from aggressive disease, early predicting recurrence and detecting metastases or predicting effectiveness of therapies. To date efforts are fragmented, based on single-institution, size-limited and vendorspecific datasets while available PCa public datasets (e.g. US TCIA) are only few hundred cases making model generalizability impossible.

The ProCAncer-I project brings together 20 partners, including PCa centers of reference, world leaders in AI and innovative SMEs, with recognized expertise in their respective domains, with the objective to design, develop and sustain a cloud based, secure European Image Infrastructure with tools and services for data handling. The platform hosts the largest collection of PCa multi-parametric (mp)MRI, anonymized image data worldwide (>17,000 cases), based on data donorship, in line with EU legislation (GDPR). Robust AI models are developed, based on novel ensemble learning methodologies, leading to vendor-specific and -neutral AI models for addressing 8 PCa clinical scenarios.

To accelerate clinical translation of PCa AI models, we focus on improving the trust of the solutions with respect to fairness, safety, explainability and reproducibility. Metrics to monitor model performance and a causal explainability functionality are developed to further increase clinical trust and inform on possible failures and errors. A roadmap for AI models certification is defined, interacting with regulatory authorities, thus contributing to a European regulatory roadmap for validating the effectiveness of AI-based models for clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

1. histological confirmed PCa or suspicion of PCa (abnormal PSA values and/or positive DRE);
2. magnetic resonance imaging examination, including at least a high-resolution axial T2-weighted imaging and axila diffusion-weighted imaging (dynamic contrast-enhanced imaging is recommended, but not mandatory);
3. age ≥ 18 years at the time of diagnosis
4. signed written informed consent form (only for prospective enrollement).

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent MRI examination with pathological confirmation of prostate cancer (positive group) or at least 1-year follow-up to exclude presence of prostate cancer (negative group).
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
To create a repository (Prostate-NET) of retrospective MRI examinations with related clinical and pathology data dedicated to prostate cancer. | 24 months
To use the retrospective data collection (Prostate-NET) to solve 9 different clinical scenarios to improve diagnosis, characterization, treatment and follow-up of men with prostate cancer. | 36 months
To develop vendor-specific and vendor neutral AI models exploiting the prospective data that will be uploaded to the Prostate-NET platform. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Manolis Tsiknakis, Study Director — FORTH; Nickolas Papanikolau, Study Chair — Fundacao Champalimaud; Kostantinos Marias, Study Chair — FORTH
Locations (1):
- Fondazione del Piemonte per l'Oncologia, Candiolo, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes